CLINICAL TRIAL: NCT01882751
Title: In Vivo Determination & Comparison of Knee Kinematics for Subjects Implanted With Either a Personalized ConforMIS or Traditional Knee Implant
Brief Title: In Vivo Comparison of Knee Kinematics for Subjects Implanted With Either a ConforMIS or Traditional Knee Implant
Status: Completed | Type: Observational
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: Komistek 2
Record Dates: First submitted 2013-05-21; First posted 2013-06-20 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Complications; Arthroplasty
Keywords: kinematics; knee joint

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- ConforMIS: Patients with ConforMIS implants
  Interventions: Device: Conformis CR Total Knee Replacement
- Standard Total Knee Implant: Patients implanted with standard total knee implant
  Interventions: Device: Off the Shelf

INTERVENTIONS:
Device: Conformis CR Total Knee Replacement — iTotal CR by Conformis
  Groups: ConforMIS
Device: Off the Shelf — A standard knee replacement not using ConforMIS' iFit technology
  Groups: Standard Total Knee Implant

SUMMARY:
A better understanding of knee joint kinematics is important to explain the premature polyethylene wear failures within total knee arthroplasties (TKAs) and to help design a prosthesis that most closely approximates the normal knee. Previously, most experimental studies of knee kinematics have involved cadaveric, in vitro analyses, or have not tested the knee in a weight-bearing mode. Others have used exoskeletal linkages and skin markers that permit error due to undesired motions between markers and the underlying bone. More recently, fluoroscopy has been used to assess in vivo kinematics for subjects having a TKA.

ConforMIS has attempted to follow a clearly different path than the major orthopaedic companies. They have chosen to offer patients a personalized knee implant based off of each patient's femoral and tibial bone geometry. The hypothesis is that these subjects will experience a more normal-like kinematic pattern, eliminating paradoxical anterior sliding during weight-bearing knee flexion. Therefore, the objective for this study is to analyze the in vivo kinematics for 25 patients implanted with a personalized ConforMIS TKA and 25 patients implanted with a traditional TKA design to determine if there are any kinematic differences between these TKA designs.

DETAILED DESCRIPTION:
Each subject will be asked to perform five activities in one continuous sequence: (1) stand up from a chair, (2) walk up stairs, (3) walk down stairs, (4) level walking, and (5) a deep knee bend. Subjects will be video recorded from the waist down while performing the activities. The speed level of each trial will be based on the comfort level of the patient. The fluoroscopic images will be stored digitally for subsequent analysis on secure servers and workstations at the University of Tennessee.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months post-op
* Between 40-70 years of age
* Body weight of less than 250lbs
* TKA patients will be judged clinically successful with an American Knee Society score of greater than 90
* Must have post-op passive flexion of 100 degrees with no ligamentous laxity or pain
* Participants must be able to walk on level ground without aids and ascend/descend stairs without assistance.
* Subjects will either a ConforMIS™ TKA or a traditional TKA manufactured by any other orthopaedic company.
* Patients must be between 160cm (5'3) and 193cm (6'4) tall.

Exclusion criteria:

* Subjects not willing to sign the Informed Consent and HIPAA forms to participate in the study
* BMI >40
* Pregnant females
* Surgical procedures conducted within the past 6 months other than TKA
* Subjects from the physician's list who do not meet study requirements
* Unwilling or unable to comply with study requirements
* Participation in another clinical study which would confound results

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are at least 6 month post-op with a ConforMIS knee replacement or a standard total knee replacement who meets the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2013-06; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Kinematic Patterns during gait | at least 6 months post surgery
  There are multiple parameters captured by fluoroscopy that will be assessed during these 4 activities including:
  1. Anterior/posterior medial and lateral condyle contact positions
  2. Axial rotation of the femoral component relative to the tibial component
  3. Condylar lift-off will be determined by measuring the distances from the medial and lateral condyles to the polyethylene insert surface
  4. Weight-bearing range-of-motion.
Kinematic patterns during deep knee bend | at least 6 months post surgery
  There are multiple parameters captured by fluoroscopy that will be assessed during these 4 activities including:
  1. Anterior/posterior medial and lateral condyle contact positions
  2. Axial rotation of the femoral component relative to the tibial component
  3. Condylar lift-off will be determined by measuring the distances from the medial and lateral condyles to the polyethylene insert surface
  4. Weight-bearing range-of-motion.
Kinematics patterns during going up and down stairs | at least 6 months post surgery
  There are multiple parameters captured by fluoroscopy that will be assessed during these 4 activities including:
  1. Anterior/posterior medial and lateral condyle contact positions
  2. Axial rotation of the femoral component relative to the tibial component
  3. Condylar lift-off will be determined by measuring the distances from the medial and lateral condyles to the polyethylene insert surface
  4. Weight-bearing range-of-motion.
Kinematics patterns during getting up from chair | at least 6 months post surgery
  There are multiple parameters captured by fluoroscopy that will be assessed during these 4 activities including:
  1. Anterior/posterior medial and lateral condyle contact positions
  2. Axial rotation of the femoral component relative to the tibial component
  3. Condylar lift-off will be determined by measuring the distances from the medial and lateral condyles to the polyethylene insert surface
  4. Weight-bearing range-of-motion.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Komistek, PhD, Principal Investigator — Univeristy of Tennessee; Harold Cates, MD, Principal Investigator — Tennessee Orthopaedic Clinics
Locations (2):
- United States (2):
  - Tennessee Orthopaedic Clinics, Knoxville, Tennessee
  - University of Tennessee, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No